CLINICAL TRIAL: NCT07308964
Title: A Comparative Study of Shortened (4-Infusion) Versus Standard (8-Infusion) Teprotumumab Regimens in Patients With Thyroid Eye Disease (TED) Exhibiting an Early Optimal Clinical Response
Brief Title: Comparison of the Efficacy and Safety of 4 vs. 8 Treatments With Tepezza (Teprotumumab) for Thyroid Eye Disease
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Principal Investigator, Prof. Landau Prat Daphna, Oculoplastic and Orbital surgeon, Sheba Medical Center
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: SMC-2514-25
Record Dates: First submitted 2025-12-28; First posted 2025-12-30 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Thyroid Eye Disease; Thyroid Eye Disease, TED; Thyroid Eye Disease (TED)
Keywords: thyroid eye disease; TED; Tepezza; Teprotumumab
MeSH Terms: conditions — Graves Ophthalmopathy | interventions — teprotumumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Standard of Care (Active Comparator): Participants in this arm will receive the full standard-of-care course of Teprotumumab. This consists of a total of 8 intravenous (IV) infusions.
  Interventions: Drug: Teprotumumab Injection [Tepezza]
- Shortened Treatment (Experimental): Participants in this arm will receive a shortened course of Teprotumumab. After demonstrating an "Early Optimal Clinical Response" following the first 4 infusions, treatment will be discontinued. These participants will receive a total of 4 intravenous (IV) infusions instead of the standard 8.
  Interventions: Drug: Teprotumumab Injection [Tepezza]

INTERVENTIONS:
Drug: Teprotumumab Injection [Tepezza] — As a standard of care Teprotumumab is administered intravenously every 3 weeks for a total of 8 infusions (24 weeks).
  In the Shortened Arm participants receive a total of 4 infusions (12 weeks) provided they met the "Early Optimal Clinical Response" criteria at Week 12.

SUMMARY:
The goal of this interventional study is to compare the clinical outcomes of shortened 4-infusion course versus the standard 8-infusion course of Teprotumumab (Tepezza) in patients with active Thyroid Eye Disease (TED).

The main question it aims to answer is:

* Is a shorter course equally effective and safe for patients who respond well early in treatment.

Participants who demonstrate an early clinical response as part of their treatment with Teprotumumab will receive a shorter protocol of 4 infusions instead of the standard 8.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have a confirmed diagnosis of active Thyroid Eye Disease (TED).
* Participants must be eligible for and have started the standard Teprotumumab (Tepezza) treatment protocol.
* Participants must demonstrate a significant clinical response by the 4th infusion.
* Ability to understand and provide signed written informed consent.

Exclusion Criteria:

* Previous use of Teprotumumab or other biologic therapies for TED.
* Participants who do not show early clinical response after the 4th infusion.
* Participants who have any medical contraindications to Teprotumumab or any of its components.
* Participants who have any known hearing problems.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2028-01 (Estimated); Study Completion 2028-05 (Estimated)

PRIMARY OUTCOMES:
Clinical Response | 1 year
  Defined as a reduction of 2 or more points in the Clinical Activity Score (CAS), improvement in diplopia and exophthalmos.